CLINICAL TRIAL: NCT02605070
Title: Pilot Study on the Effects of FSH Treatment on the Epigenetic Characteristics of Spermatozoa in Infertile Patients With Severe Oligozoospermia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: UNDER RECRUITMENT
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSH_IMEN
Record Dates: First submitted 2015-11-09; First posted 2015-11-16 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2017-05

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Urofollitropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infertility group (Experimental): Patients referred will be evaluated to participate in the study and then asked to take part.In this visit,the normal protocol for infertility patients will be followed and at least 2 spermiograms and a blood test analyzing the following parameters:FSH, LH,Estradiol,Total testosterone,SHBG, Albumin,Calculation of bioavailable testosterone,Prolactin.If these tests have not been performed,a second baseline visit will be scheduled.Should the patient meet all the inclusion criteria and after the patient has signed an informed consent form agreeing to participate in the study,the physician will prescribe the medication and schedule visits.Before initiating the treatment, they will provide a semen sample.This sample will be sent to the Center for Reproductive Biology,where the sample will be subjected to epigenetic analysis.The patient will be given samples of Bravelle.It is administered subcutaneously.The dose will be 150 IU 3times a week for 3months
  Interventions: Drug: Bravelle
- Fertily group (No Intervention): Patients who volunteer will be informed of the nature of the study and asked to sign the informed consent form. At least two spermiograms will be performed along with a blood test analyzing the following parameters:FSH,LH,Estradiol,Total testosterone,SHBG,Albumin,Estimation of bioavailable testosterone,Prolactin.
  A second baseline visit will be scheduled to evaluate the test results and to check whether these subjects meet all the inclusion criteria for the control group. Those subjects will provide a semen sample which will be stored at -20º C.
  Outpatient visit: week twelve: a physical exam will be carried out to identify any adverse reactions. A blood test and a semen sample will also be obtained.

INTERVENTIONS:
Drug: Bravelle — Bravelle will be provided to all patients in the treatment group by the principal investigator (PI) or another member of the research team.
  From week nine on, the patients will undergo a physical examination on three different occasions to assess the appearance of any adverse reactions during treatment. It will be up to the patient to communicate the appearance of signs or symptoms which could be associated with the use of the drug.
  At week 12 the patient will be scheduled for another visit to perform a semen study and to measure new hormone levels. To this end, a blood test will be carried out (FSH, LH, estradiol, total testosterone, SHBG, and albumin to calculate the amount of bioavailable testosterone). A semen sample will also be obtained to carry out a spermiogram according to WHO guidelines; part of this sample will be used for epigenetic analysis.
  Arms: Infertility group

SUMMARY:
Single center, prospective, open clinical study to determine the genomic imprint (epigenetic modification) in a series of male infertility patients with alterations in their spermiogram (oligozoospermia) compared to a group of fertile patients in order to evaluate the effect of FSH ( follicle stimulating hormone) administration on these modifications and on male infertility.

DETAILED DESCRIPTION:
Single center, prospective, open clinical study to determine the genomic imprint (epigenetic modification) in a series of male infertility patients with alterations in their spermiogram (oligozoospermia) compared to a group of fertile patients in order to evaluate the effect of FSH ( follicle stimulating hormone) administration on these modifications and on male infertility.

Main objective: To determine the genomic imprint (epigenetic modification) in a series of male infertility patients with alterations in their spermiogram (oligozoospermia) compared to a group of fertile patients in order to evaluate the effect of FSH administration on these modifications and on male infertility.

Secondary objectives

* To assess the main characteristics of the spermiograms of infertility patients before and after FSH treatment.
* To assess modifications in the hormones involved in sperm formation in infertility patients before and after treatment.
* To analyze the results of assisted reproduction treatments in patients receiving FSH treatment.

ELIGIBILITY:
* Inclusion criteria for the infertility treatment group (n=30)

  1. Between 25-45 years of age.
  2. Total sperm concentration (concentration in millions/mL x volume in mL) between 1-10 million (oligozoospermia) in at least 2 spermiograms obtained after a 2-4 day period of sexual abstinence and with a 7-day separation period between tests.
  3. Caucasian.
  4. Inability of the couple to become pregnant after one year of sexual relations without using any type of contraception.
  5. FSH 2-12 IU/mL.
  6. Total testosterone >300 ng/mL and bioavailable testosterone (calculated with the Sexual Hormone Binding Globulin or SHBG albumin) >145 ng/dL.
* Inclusion criteria for the control group of fertile males (n=15)

  1. Between 25-45 years of age.
  2. Caucasian.
  3. Sperm concentration and motility above the 5th percentile according to the parameters set forth in the 5th edition of the World Health Organization (WHO) guidelines in at least two spermiograms obtained after a 2-4 day period of sexual abstinence and with a 7-day period between tests.
  4. Seminal volume >1 mL.
  5. Estradiol <50 pg/mL
  6. FSH <4.5 IU/L.
  7. Total testosterone >300 ng/dL and bioavailable testosterone >145 ng/dL.
  8. No vasectomy.
  9. Has sired a child within the past 5 years.
* Exclusion criteria for the infertility treatment group.

  1. Total sperm concentration <1 million.
  2. Sperm motility of 0%.
  3. History of cryptorchidism, malignant or benign tumors, known chromosomal abnormalities, testicular tor- sion, testicular trauma, orchitis.
  4. Drug use in the past 120 days. thyroid dysfunction
  5. Medical history:thyroid dysfunction, blood disease, diabetes.
  6. Use of anabolic steroids in the past 2 years or for more than 2 years.
  7. Body mass index >30 kg/m .
  8. Intake of over 21 units of alcohol/week in the past 120 days.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Epigenetic modification | 12 weeks after treatment.
  To determine the genomic imprint (epigenetic modification) in a series of male infertility patients with alterations in their spermiogram (oligozoospermia) compared to a group of fertile patients in order to evaluate the effect of FSH administration on these modifications and on male infertility

SECONDARY OUTCOMES:
To assess the main characteristics of the spermiograms of infertility patients before and after FSH treatment. | First week and end of treatment visit (12 weeks).
  To assess the main characteristics of the spermiograms of infertility patients before and after FSH treatment.
To assess modifications in the hormones involved in sperm formation in infertility patients before and after treatment. | First week and end of treatment visit (12 weeks)
  To assess modifications in the hormones involved in sperm formation in infertility patients before and after treatment.
Pregnancy rate. | 6-7 weeks after transfer of the embryo.
  To analyze the results of assisted reproduction treatments in patients receiving FSH treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari i Politècnic La Fe, Valencia, Spain

REFERENCES:
- [Result] Boivin J, Bunting L, Collins JA, Nygren KG. International estimates of infertility prevalence and treatment-seeking: potential need and demand for infertility medical care. Hum Reprod. 2007 Jun;22(6):1506-12. doi: 10.1093/humrep/dem046. Epub 2007 Mar 21. PMID 17376819
- [Result] Dohle GR, Halley DJ, Van Hemel JO, van den Ouwel AM, Pieters MH, Weber RF, Govaerts LC. Genetic risk factors in infertile men with severe oligozoospermia and azoospermia. Hum Reprod. 2002 Jan;17(1):13-6. doi: 10.1093/humrep/17.1.13. PMID 11756355
- [Result] Simoni M, Gromoll J, Dworniczak B, Rolf C, Abshagen K, Kamischke A, Carani C, Meschede D, Behre HM, Horst J, Nieschlag E. Screening for deletions of the Y chromosome involving the DAZ (Deleted in AZoospermia) gene in azoospermia and severe oligozoospermia. Fertil Steril. 1997 Mar;67(3):542-7. doi: 10.1016/s0015-0282(97)80083-0. PMID 9091344
- [Result] Gianotten J, Lombardi MP, Zwinderman AH, Lilford RJ, van der Veen F. Idiopathic impaired spermatogenesis: genetic epidemiology is unlikely to provide a short-cut to better understanding. Hum Reprod Update. 2004 Nov-Dec;10(6):533-9. doi: 10.1093/humupd/dmh045. Epub 2004 Oct 1. PMID 15465836
- [Result] Jenkins TG, Carrell DT. Dynamic alterations in the paternal epigenetic landscape following fertilization. Front Genet. 2012 Jul 31;3:143. doi: 10.3389/fgene.2012.00143. eCollection 2012. PMID 23024648
- [Result] Kelly TL, Li E, Trasler JM. 5-aza-2'-deoxycytidine induces alterations in murine spermatogenesis and pregnancy outcome. J Androl. 2003 Nov-Dec;24(6):822-30. doi: 10.1002/j.1939-4640.2003.tb03133.x. PMID 14581508
- [Result] Houshdaran S, Cortessis VK, Siegmund K, Yang A, Laird PW, Sokol RZ. Widespread epigenetic abnormalities suggest a broad DNA methylation erasure defect in abnormal human sperm. PLoS One. 2007 Dec 12;2(12):e1289. doi: 10.1371/journal.pone.0001289. PMID 18074014
- [Result] Kobayashi H, Sato A, Otsu E, Hiura H, Tomatsu C, Utsunomiya T, Sasaki H, Yaegashi N, Arima T. Aberrant DNA methylation of imprinted loci in sperm from oligospermic patients. Hum Mol Genet. 2007 Nov 1;16(21):2542-51. doi: 10.1093/hmg/ddm187. Epub 2007 Jul 17. PMID 17636251
- [Result] Benchaib M, Braun V, Ressnikof D, Lornage J, Durand P, Niveleau A, Guerin JF. Influence of global sperm DNA methylation on IVF results. Hum Reprod. 2005 Mar;20(3):768-73. doi: 10.1093/humrep/deh684. Epub 2005 Jan 7. PMID 15640258
- [Result] Reyes-Fuentes A, Chavarria ME, Carrera A, Aguilera G, Rosado A, Samojlik E, Iranmanesh A, Veldhuis JD. Alterations in pulsatile luteinizing hormone and follicle-stimulating hormone secretion in idiopathic oligoasthenospermic men: assessment by deconvolution analysis--a clinical research center study. J Clin Endocrinol Metab. 1996 Feb;81(2):524-9. doi: 10.1210/jcem.81.2.8636262.
- [Result] Fujisawa M, Kanzaki M, Hayashi A, Tanaka H, Okada H, Arakawa S, Kamidono S. Alteration of the hypothalamus-pituitary-testis axis in oligozoospermic men with normal gonadotropin levels. Int J Urol. 1995 Sep;2(4):273-6. doi: 10.1111/j.1442-2042.1995.tb00471.x. PMID 8564748
- [Result] Boissonnas CC, Jouannet P, Jammes H. Epigenetic disorders and male subfertility. Fertil Steril. 2013 Mar 1;99(3):624-31. doi: 10.1016/j.fertnstert.2013.01.124. PMID 23714437